CLINICAL TRIAL: NCT06929494
Title: Candidemia in Critically Ill Patients: Risk Factors and Predictive Factors
Brief Title: Candidemia in Critically Ill Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: MMC-0086-25
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Identification of risk factors for candidemia — Identification of risk factors for candidemia

SUMMARY:
Candidal sepsis (candidemia) is a criticals problem in patients hospitalized in the intensive care unit, with a significant impact on morbidity and mortality. Risk factors for candidemia in intensive care patients included age, presence of a central venous catheter, inpatient surgery, and administration of parenteral nutrition (TPN). Mortality in patients with candidemia is estimated at 50-60%. Early identification and treatment, including control of the source of infection, are essential to improve morbidity and mortality in these patients.

In this study, we would like to identify risk factors for the development of candidemia in intensive care patients, including those who have not undergone abdominal surgery, and to examine what percentage of patients who developed candidemia were given empirical antifungal therapy and what factors influenced the decision to give or not to give such empirical therapy.

Study design: A retrospective study based on data collection from computerized systems will include patients who were hospitalized in the intensive care unit from January 2014 to December 2024 and were diagnosed with Candida in at least one blood culture.

ELIGIBILITY:
Inclusion Criteria: Patients admitted to the ICU from January 2014 to December 2024 and had at least one positive blood culture for candidemia -

Exclusion Criteria: Missing data

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU from January 2014 to December 2024 and had at least one positive blood culture for candidemia
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Identification of risk factors for candidemia | Throughout ICU stay (from admission to 28 days post ICU discharge)
  Identification of risk factors for candidemia

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No